CLINICAL TRIAL: NCT01421030
Title: Outcomes in Patients and Their Closest Relatives Treated for Congenital Heart Disease With Catheter Based or Surgical Techniques.
Acronym: MEQC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Brith Andresen, CNS, MNSc, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011/210
Record Dates: First submitted 2011-06-24; First posted 2011-08-22 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Congenital Heart Defects
Keywords: quality of life; congenital heart disease; open heart surgery; percutaneous pulmonary valve implantation; costs
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- quality of life, clinical outcomes and costs (Other): Quality of life, clinical outcomes and costs after two different treatment options in patients and closest relatives
  Interventions: Procedure: Percutaneous pulmonary valve implantation or open heart surgery

INTERVENTIONS:
Procedure: Percutaneous pulmonary valve implantation or open heart surgery — Outcomes before percutaneous pulmonary valve implantation or open heart surgery before, 1, 3, 6 and 12 months after the treatment

SUMMARY:
This study compares clinical, self- reported and cost outcomes in children and adolescents treated with pulmonary valve implantation, percutaneous versus open surgical technique. Since cardiac surgery in children and adolescents affect the whole family, the experience of the patients and their closest relatives are recorded and analysed separately. Cost may be an important factor in the choice of technology (1). Hence, the present study also aims to compare savings in costs, percutaneous versus open technique, related to the individual, their family and society.

1.2 Research questions

1. Percutaneous pulmonary valve implantation or open heart surgery; what are the patients' and their closest relatives narrative experiences
2. Is there a difference in patient and their closest relatives reported outcomes, measured as health related quality of life, in patients with congenital pulmonary disease before the event, 1, 3, 6 and 12 months after percutaneous intervention versus open heart surgery approach?
3. What is the relationship between patient reported outcomes and clinical outcomes before, 1, 3, 6 and 12 months after the treatment?
4. Are there savings in costs related to the individual and their family and society between the two techniques?

ELIGIBILITY:
Inclusion Criteria:

* secure indication of pulmonary valve dysfunction (stenosis and, or regurgitation)
* an indication of surgical correction
* body weight according to the recommendation from the producer of the device
* moderate to serious dilatation of right ventricle
* considerable leak in the tricuspidal valve
* information from former surgery; conduit size, gradient of the stenosis measured by EKKO/MR/ catheterization, X-ray.
* be able to speak and communicate well in Norwegian.

Exclusion Criteria:

* aggressive endocarditis
* not circumferential deposit of calcium
* < 20 kg
* not able to understand, speak or communicate well in Norwegian

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life | up to 12 month's after treatment
  Percutaneous pulmonary valve implantation or open heart surgery; what are the patients and their closest relatives narrative experiences. Measured before the event, 1, 3, 6, and 12 month's after treatment.

SECONDARY OUTCOMES:
Clinical outcomes | up to 12 months after treatment
  What is the relationship between patient reported outcomes and clinical outcomes before, 1, 3, 6 and 12 months after the treatment
  Is there a difference in the effect of percutaneous versus open surgical technique on operative time, complication rate and reoperations in the peri- and postoperative period?
Are there savings in costs related to the individual and their family and society between the two techniques? | up to 12 months after surgery
  In order to describe and compare the differences in costs with patients outcomes and quality-adjusted life years, this study aim to calculate both in-hospital care and out-patient clinical costs between percutaneous pulmonary valve implantation and conventional open heart surgery. Measured Before the event, 1, 3, 6 and 12 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, Professor/Head of Department, Principal Investigator — The Interventional Centre, Rikshospitalet, Oslo University Hospital
Locations (1):
- The Interventional Centre, Rikshospitalet, Oslo University Hospital, Oslo, Sognsvannsvn 20, Norway